CLINICAL TRIAL: NCT06593405
Title: The Role of Occupational Therapy for Improving Medication Management for Persons With AMD, Diabetic Retinopathy (DR) and Glaucoma
Brief Title: The Role of Occupational Therapy for Improving Medication Management for Persons With AMD, DR and Glaucoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: MCPHS University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-2024-84
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-04

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study to determine outcomes with occupational therapy (OT) medication management interventions/strategies for persons with Age-related Macular Degeneration (AMD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving OT interventions (Experimental): All participants will receive all OT interventions
  Interventions: Combination Product: occupational therapy interventions for low vision care

INTERVENTIONS:
Combination Product: occupational therapy interventions for low vision care — Occupational therapists utilize many different treatment strategies when caring for the client with low vision. Oftentimes, the client is unaware of these strategies which may improve occupational performance during a valued activity. Interventions include task lighting, organizational strategies, smart apps, contrast, enlarged print, typoscopes and electronic magnification devices.

SUMMARY:
The goal of this clinical trial is to learn if education about additional task lighting, enhanced contrast, enlarged print instructions, smart apps and organizational strategies will improve medication management skills. The main questions it aims to answer are:

Does additional task lighting, enhanced contrast, enlarged print instructions, smart apps and organizational strategies improve medication management skills, reduce errors and improve functional use of remaining vision for this task?

Participants will:

Oftentimes, the client is unaware of these strategies which may improve occupational performance during a valued activity. Clients with AMD, DR or Glaucoma who choose to receive the one hour OT service will be provided with 1:1 education regarding the devices and strategies that may improve their ability to perform medication management skills.

DETAILED DESCRIPTION:
Many clients with low vision are unaware of OT, or the services OT can provide to assist with low vision needs. Clients with AMD, DR or Glaucoma who choose to receive the one hour OT service will be provided with 1:1 education regarding the devices and strategies that may improve their ability to perform medication management skills. Clients will complete the MediCog and the Revised-Self-Report Assessment of Functional Visual Performance (R-SRAFVP) assessment tools with the assistance of the OT. These tools will inform the therapist to areas of client needs and allow for focus on intervention to support these challenges. Follow up in OT 4 weeks post intervention will allow therapist to reassess the effectiveness of interventions provided via a phone or in-person interview as well as provide the assessments again. Second set of data from these assessments will be compared to initial findings obtained.

ELIGIBILITY:
Inclusion Criteria:

* Clients with AMD, DR or Glaucoma
* Clients who choose to participate will allow their deidentified data to be evaluated for outcomes.

Exclusion Criteria:

* Clients with other age related eye diseases other than AMD, DR or Glaucoma.
* Clients who do not wish to participate in this study.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Revised Self Report Assessment of Functional Visual | Results from the Revised-Self-Report Assessment of Functional Visual Performance assessment will be determined on day 1 and 4 weeks later
  A standardized assessment which provides information on how well adults with vision loss can perform daily tasks. This tool has 33 assessment components and a higher score indicates less functional impairment. A lower score indicates a higher impairment.
MediCog Screening Tool | Results from the MediCog will be determined on day 1 and will be obtained 4 weeks later
  The Medi-Cog has a maximum score of 10 points, and a score of 7 or lower may indicate cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dowling, OTD, Principal Investigator — MCPHS University
Locations (1):
- MCPHS 10 Lincoln Square, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be analyzed and results will be shared in the form of publication in a peer reviewed journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication

REFERENCES:
- [Background] Occupational Therapy's Role in Medication Management. Am J Occup Ther. 2017 Nov/Dec;71(Supplement_2):7112410025p1-7112410025p20. doi: 10.5014/ajot.2017.716S02. No abstract available. PMID 29309002
- See also: American Occupational Therapy Association link to professional information — https://www.aota.org/publications/ot-practice/ot-practice-issues/2020/medication-adherence